CLINICAL TRIAL: NCT05322031
Title: The Impact of Aripiprazole Long-acting on Myelin and Cognition in the Onset of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARIANNA
Record Dates: First submitted 2022-03-16; First posted 2022-04-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia; Myelin Degeneration; Cognition Disorder
Keywords: Onset of schizophrenia; Aripiprazole long-acting; Myelin; Cognition
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Onset of depression (Experimental): 15 participants with onset of schizophrenia who, after a period of stabilization with aripiprazole in oral formulation, would begin therapy with long-acting aripiprazole, or already in therapy with long-acting aripiprazole since no more than two weeks.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Patiens who underwent a a period of stabilization with aripiprazole in oral formulation that begin therapy with long-acting aripiprazole, or already in therapy with long-acting aripiprazole from no more than two weeks.
  Other Names: Abilify Maintena; Long-acting aripiprazole

SUMMARY:
The general objective of this interventional study is to explore the impact of long-acting arpiprazole on brain structure, in particular potential neurotrophic effects, neurogenetic and neuroprotective that could counteract the progressive neuronal degeneration inherent in the schizophrenic pathology itself.

Each subject will undergo a structured clinical interview to assess the presence/absence of Axis I psychiatric disorders (SCID-5 CV). This evaluation is carried out in common clinical practice as a tool to support diagnosis in patients with suspected schizophrenia.

In all subjects, the cognitive profile will be evaluated through the Brief Assessment of Cognition in schizophrenia (BAC-S). The degree of psychotic symptomatology reported through the administration of specific psychopathological scales such as the Brief Psychiatric Rating Scale (BPRS) and the Positive and Negative Syndrome Scale (PANSS) will also be measured. Further clinical data will be extrapolated from medical records and interviews with psychiatrists, if available.

In patients diagnosed with schizophrenia at the first psychotic episode, the administration of pharmacological therapy with long-acting aripiprazole will take place following the indications of the relevant data sheet.

At the U.O.C. of Neuroradiology of the Fondazione, all enrolled subjects will undergo a 3-Tesla multimodal neuroimaging session that includes:

* T1-weighted sequences: to study the volumetric differences of white and grey matter between subjects before and after treatment;
* Acquisition of myelin sequences: to assess the differences in myelin between subjects before and after treatment;
* DTI sequences: to assess differences in white matter bundles between subjects before and after treatment.

The degree of psychotic symptomatology reported will be evaluated by the repetition of psychopathological scales (BPRS, PANSS). Three months after the start of therapy all patients who have joined the study will carry out a 3T NMR of extra standard care control.

DETAILED DESCRIPTION:
The general objective of this interventional study is to explore the impact of long-acting arpiprazole on brain structure, in particular potential neurotrophic effects, neurogenetic and neuroprotective that could counteract the progressive neuronal degeneration inherent in the schizophrenic pathology itself. In other words, the primary objective is to assess if the achievement of therapeutic control of the pathology through the use of antipsychotic drug corresponds to a change in the brain structure, both in terms of morphology and connectivity. A further objective will be to evaluate the effect of long-acting aripiprazole on the clinical outcome (in terms of relapses and clinical symptoms), on the overall functioning and cognitive performance of patients at the first psychotic episode in the context of a diagnosis of schizophrenia. The study will be attended by patients with onset of schizophrenia recruited from the Psychiatric Service of Diagnosis and Care and the Day Hospital of the U.O.C. of Psychiatry of the IRCCS Fondazione Ca' Granda, Ospedale Maggiore Policlinico in Milan. A team of psychologists and medical experts of the UOC of Psychiatry of the Fondazione will conduct the process of enrollment and participation in the study. Each subject will undergo a structured clinical interview to assess the presence/absence of Axis I psychiatric disorders (SCID-5 CV). This evaluation is carried out in common clinical practice as a tool to support diagnosis in patients with suspected schizophrenia.

In all subjects, the cognitive profile will be evaluated through the Brief Assessment of Cognition in schizophrenia (BAC-S). In patients, the degree of psychotic symptomatology reported through the administration of specific psychopathological scales such as the Brief Psychiatric Rating Scale (BPRS) and the Positive and Negative Syndrome Scale (PANSS) will also be measured. Further clinical data will be extrapolated from medical records and interviews with psychiatrists, if available.

In patients diagnosed with schizophrenia at the first psychotic episode, the administration of pharmacological therapy with long-acting aripiprazole will take place following the indications of the relevant data sheet, upon prescription of the doctor, on the basis of the clinical assessment and independently of participation in the study. The introduction of aripiprazole long-acting drug therapy will follow a period of stabilization with oral aripiprazole, as reported in the data sheet.

At the U.O.C. Neuroradiology of the Fondazione, all enrolled subjects will undergo a 3-Tesla multimodal neuroimaging session that includes:

* T1-weighted sequences: to study the volumetric differences of white and grey matter between subjects before and after treatment;
* Acquisition of myelin sequences: to assess the differences in myelin between subjects before and after treatment;
* DTI sequences: to assess differences in white matter bundles between subjects before and after treatment.

This resonance is an ordinary clinical practice for patients with psychosis. It is important to note that 3T MRI is no longer considered high-field and is now commonly used in the regular clinical practice.

For patients, clinical reassessment visits (one per month for 3 months) are already scheduled by practice for the normal management of the clinical situation. The degree of psychotic symptomatology reported will be evaluated by the repetition of psychopathological scales (BPRS, PANSS). Three months after the start of therapy all patients who have joined the study will carry out a 3T NMR of extra standard care control.

ELIGIBILITY:
Inclusion Criteria:

* onset of schizophrenia diagnosed by the support of structured clinical interview (SCID-5 CV) by specialized medical staff;
* age 18 to 65 years, who, after a period of stabilization with aripiprazole in oral formulation, must start a therapy with long-acting aripiprazole for clinical needs (and therefore regardless of participation in the study) or already in therapy with long-acting aripiprazole not more than two weeks;
* absence of other psychotropic drugs for at least two weeks prior to the start of the study;
* to have signed the informed consent to participate in the study;
* for women of child-bearing age, a pregnancy test (betaHCG urine or blood test) must be carried out immediately before the start of therapy and a highly effective method of contraception must be taken for the duration of the treatment.

Exclusion Criteria:

* presence of codiagnosis with other psychiatric (based on SCID-5 CV) or neurological pathologies;
* previous antipsychotic therapies. Patients previously stabilized with other antipsychotic drugs will still be admitted, provided that they are taken for a period of time not exceeding one month and provided that they have not been taken within 2 weeks prior to enrollment, except for aripiprazole in oral formulation, the intake of which is necessary for the inclusion of aripiprazole in long-acting formulation.
* contraindications to taking aripiprazole long-acting as per SPC;
* history of intellectual disability;
* abuse of alcohol or substances during the preceding six months;
* presence of absolute or relative contraindications to the execution of MRI;
* underage patients;
* pregnant women (if the pregnancy occurs during the study, the patient will be excluded from the continuation of the study) or women who have not performed a pregnancy test negative result before the start of therapy and who do not adopt valid contraceptive methods.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Brain structural modifications in terms of myelination of the white matter measured using magnetic resonance imaging | 3 months of therapy
  Evaluation of the modification of the myelination of white matter bundles (in terms of Myelin Water Fraction - MWF) after antipsychotic therapy with aripiprazole long-acting compared to baseline measured using magnetic resonance imaging.

SECONDARY OUTCOMES:
Evaluation of efficacy as assessed by Positive and Negative Syndrome scale | 3 months from baseline.
  Evaluation of the efficacy of aripiprazole long-acting on the clinical outcome, measured by variation of the score of the psychopathological PANSS (Positive and Negative Syndrome Scale) scale with respect to the baseline.
Evaluation of efficacy as assessed by Brief Psychiatric Rating Scale | 3 months from baseline.
  Evaluation of the efficacy of aripiprazole long-acting on the clinical outcome, measured by variation of the score of the psychopathological BPRS (Brief Psychiatric Rating Scale) scale with respect to the baseline.
Changes in cognitive performance through Brief Assessment of Cognition in schizophrenia scale | 3 months from baseline.
  Evaluation of the efficacy of aripiprazole long-acting on the cognitive performance, measured in terms of variations of neuropsychological BAC-S (Brief Assessment of Cognition in schizophrenia) scale scores with respect to the baseline
Number of adverse and toxic events due to the administration of aripiprazole | Through study completion (1 year)
  Evaluation of serious and non-serious adverse and toxic events due to the administration of aripiprazole.
Evaluation of the statistical correlation between plasma levels of aripiprazole and clinical and structural assestment | Through study completion (1 year)
  Assessment of the plasma levels over time of the drug to identify a possible statistical correlation with the clinical response (in terms of changes with respect to the baseline in PANSS - Positive and Negative Syndrome Scale, BAC-S - Brief Assessment of Cognition in schizophrenia and BPRS - Brief Psychiatric Rating Scale) and with the changes in brain structure (in terms of gray matter volumes, superficial cortical area and cortical thickness) and in the myelination of white matter bundles (in terms of Myelin Water Fraction - MWF).
Changes in gray matter volumes | 3 months from baseline
  Evaluation of changes in brain structure using MRI in terms of gray matter volumes after antipsychotic therapy with long-acting aripiprazole.
Changes in superficial cortical area | 3 months from baseline
  Evaluation of changes in brain structure using MRI in terms of superficial cortical area after antipsychotic therapy with long-acting aripiprazole.
Changes in cortical thickness | 3 months from baseline
  Evaluation of changes in brain structure using MRI in terms of cortical thickness after antipsychotic therapy with long-acting aripiprazole.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Brambilla, Professor, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Massimo C Mauri, Professor, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Prof. Paolo Brambilla, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No